CLINICAL TRIAL: NCT02219451
Title: Exercise Training Improves Oscillatory Pattern and Arterial Baroreflex Control of Sympathetic Nerve Activity in Patients With Chronic Heart Failure
Brief Title: Exercise Improve Sympathetic Modulation in Chronic Heart Failure Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Raphaela Vilar Ramalho Groehs, PhD student, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: sympathetic modulation
Record Dates: First submitted 2014-08-04; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Heart Failure
Keywords: Chronic heart failure; exercise training; Sympathetic modulation; arterial baroreflex control
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise training (Experimental): We studied twenty-six chronic heart failure outpatients and they were assigned to 2 groups: Untrained (n=13) and trained (n=13).
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — exercise training

SUMMARY:
The purpose of this study is to verify the effects of exercise training on sympathetic modulation and arterial baroreflex control in patients with chronic heart failure.

DETAILED DESCRIPTION:
Retrospective study. Patients were recruited by database from Rehabilitation Unit of Cardiovascular Rehabilitation and Exercise Physiology of the Heart Institute (InCor). The aim of this study is to assess the effects of exercise training on sympathetic modulation and arterial baroreflex control in patients with chronic heart failure. The investigators studied twenty-six chronic heart failure outpatients, age 30 to 70 years, functional class II to III of New York Heart Association, left ventricular ejection fraction (LVEF) ≤40% and peak oxygen uptake (VO2) ≤20. The exclusion criteria were recent myocardial infarction or unstable angina (<3 months), heart failure duration (<3 months), permanent pacemaker dependence, atrial fibrillation, skeletal muscle abnormality (e.g., arthritis) and participation in a regular exercise program. They were assigned to 2 groups: Untrained (n=13) and trained (n=13).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure
* Age 30 to 70 years
* Functional class II to III of New York Heart Association
* Left ventricular ejection fraction (LVEF) ≤40%
* Peak oxygen uptake (VO2) ≤20

Exclusion Criteria:

* Recent myocardial infarction or unstable angina (<3 months)
* heart failure duration (<3 months)
* Permanent pacemaker dependence
* Atrial fibrillation
* Skeletal muscle abnormality (e.g., arthritis)
* Participation in a regular exercise program

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Autonomic control | 4 months
  To asses the effects of exercise training on sympathetic modulation by analyze of autonomic control in chronic heart failure patients after 4 months protocol.Time series of muscle sympathetic nerve activity and systolic arterial pressure were analyzed by autoregressive spectral analysis

SECONDARY OUTCOMES:
Arterial baroreflex control | 4 months
  To asses the effects of exercise training on arterial baroreflex by analyze of arterial baroreflex control in chronic heart failure patients after 4 months. The arterial baroreflex control was analyzed by bivariate autoregressive.

CONTACTS AND LOCATIONS:
Overall Officials: Heart Institute HC/FMUSP, HC/FMUSP, Principal Investigator — Heart Institute, University of Sao Paulo
Locations (1):
- Instituto do Coração - HC/FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Groehs RV, Toschi-Dias E, Antunes-Correa LM, Trevizan PF, Rondon MU, Oliveira P, Alves MJ, Almeida DR, Middlekauff HR, Negrao CE. Exercise training prevents the deterioration in the arterial baroreflex control of sympathetic nerve activity in chronic heart failure patients. Am J Physiol Heart Circ Physiol. 2015 May 1;308(9):H1096-102. doi: 10.1152/ajpheart.00723.2014. Epub 2015 Mar 6. PMID 25747752